CLINICAL TRIAL: NCT00164047
Title: Evaluation of Nitrous Oxide In the Gas Mixture for Anaesthesia: a Randomised Controlled Trial
Brief Title: ENIGMA - Evaluation of Nitrous Oxide In the Gas Mixture for Anaesthesia: a Randomised Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other); Australia: Theapeutic Goods Administration (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 204/02; NHMRC 236956
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2009-07

CONDITIONS: Quality of Recovery From Anaesthesia; Effects of Nitrous Oxide Following Anaesthesia; Induced Endothelial Dysfunction
Keywords: Nitrous Oxide; Anaesthesia; Anesthesia; Recovery; Quality
MeSH Terms: interventions — Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide

SUMMARY:
We aim to investigate the effectiveness and safety of nitrous oxide (N2O) in anaesthesia.

Hypothesis In patients undergoing anaesthesia for major surgery, avoidance of N2O will reduce hospital length of stay when compared with otherwise identically managed surgical patients receiving N2O as a component of their anaesthesia.

DETAILED DESCRIPTION:
There are some compelling reasons to question the routine use of nitrous oxide (N2O), also known as "laughing gas". Despite being the first anaesthetic drug introduced, and still widely used, there is sufficient doubt as to the risk-benefit profile.

There is strong evidence that N2O is a major risk factor for postoperative nausea and vomiting. It is clear that (even) brief exposure to N2O impairs methionine synthetase, an enzyme required for DNA production, red and white blood cell formation. Tissue hypoxia may be more common. These adverse effects are enhanced in "sick" patients (ie. those at highest risk, increased hospital length of stay and healthcare expenditure), and will be more likely in longer surgery. The extent of wound infection and cardiac morbidity associated with N2O is not known.

Large outcome trial data are lacking. When considering its widespread use in about 90% of all surgery around the world, small differences in outcome would have major implications for healthcare delivery. A large randomised controlled trial is necessary to answer this question.

We have recruited 2000 patients from about 25 centres around the world (mostly Australasia), who are undergoing major surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age 18 years and over
2. Planned general anaesthesia for surgery that includes a skin incision and expected to exceed two hours, and the patient is expected to be in hospital for at least three days

Exclusion Criteria:

1. Endoscopic or radiological procedures
2. Cardiac surgery
3. Marked impairment of gas-exchange (requiring Fi02> 0.3)
4. Thoracic surgery requiring one-lung ventilation (requiring Fi02> 0.3)
5. Specific circumstances where N2O is contraindicated (eg. volvulus, pulmonary hypertension, raised intracranial pressure)
6. Lack of provision of N2O.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2070 (Estimated)
Dates: Start 2003-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is hospital length of stay (LOS), defined from the start of surgery until actual hospital discharge. Patients transferred to another hospital will be tracked until final discharge to home (or other final destination). LOS is likely

SECONDARY OUTCOMES:
Secondary endpoints will be detected by a research assistant who will be masked to Group identity, using chart review up to 30 days postoperatively; confirmation of each will be sought by an independent member of the Endpoint Committee:
Wound infection - if associated with purulent discharge or a positive microbial culture (46)
Myocardial infarction - confirmed by ECG and/or troponin or CK-MB enzyme rise
Venous thromboembolism - symptomatic DVT or PE, confirmed by venography, duplex ultrasonography, V-Q scan or spiral CT, or autopsy
Stroke - a new neurological deficit persisting for 24 hours, confirmed by neurologist assessment and/or CT scan or MRI
Awareness - postoperative recollection of intraoperative events
Blood transfusion - any red cell transfusion within 30 days of surgery
Pneumothorax, atelectasis, or pneumonia - confirmed by chest x-ray; for pneumonia: also 2 or more of temp> 38oC, white cell count >12,000/ml, positive sputum culture
Severe vomiting - at least 2 episodes >6 hrs apart, or if requiring >2 doses of antiemetic medication
Quality of recovery on the morning after surgery -using the validated QoR Score instrument (14), a 9-item patient-orientated measure of early postoperative health status. This is associated with patient satisfaction.
30-day mortality - for safety analysis only (study not powered for this rare event).

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Myles, MB BS MPH MD, Principal Investigator — The Alfred
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Myles PS, Leslie K, Silbert B, Paech MJ, Peyton P. A review of the risks and benefits of nitrous oxide in current anaesthetic practice. Anaesth Intensive Care. 2004 Apr;32(2):165-72. doi: 10.1177/0310057X0403200202. No abstract available. PMID 15957712
- [Result] Myles PS, Leslie K, Chan MT, Forbes A, Paech MJ, Peyton P, Silbert BS, Pascoe E; ENIGMA Trial Group. Avoidance of nitrous oxide for patients undergoing major surgery: a randomized controlled trial. Anesthesiology. 2007 Aug;107(2):221-31. doi: 10.1097/01.anes.0000270723.30772.da. PMID 17667565
- [Derived] Leslie K, Myles PS, Chan MT, Paech MJ, Peyton P, Forbes A, McKenzie D; ENIGMA Trial Group. Risk factors for severe postoperative nausea and vomiting in a randomized trial of nitrous oxide-based vs nitrous oxide-free anaesthesia. Br J Anaesth. 2008 Oct;101(4):498-505. doi: 10.1093/bja/aen230. Epub 2008 Aug 5. PMID 18682411